CLINICAL TRIAL: NCT04567394
Title: Treating Young Adult Cannabis Use Disorder with Text Message-Delivered Peer Network Counseling
Brief Title: Cannabis Use Disorder Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: Colorado State University (Other)
Responsible Party: Principal Investigator, Michael Mason, Principal Investigator, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01DA044206-01A1 (NIH)
Record Dates: First submitted 2020-09-21; First posted 2020-09-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-05

CONDITIONS: Cannabis Use Disorder, Mild; Cannabis Use Disorder, Moderate; Cannabis Use Disorder, Severe
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Participants are randomized 1:1 to the intervention or waitlist control. Participants who complete the 6 months of waitlist control will then have the opportunity to receive the intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants randomized to the Intervention group will complete questionnaires at baseline, 1 month, 3 months, and 6 months and will receive 4 weeks of the PNC-txt intervention.
  Interventions: Behavioral: Peer Network Counseling-txt
- Waitlist Control (No Intervention): Participants randomized to the waitlist control group will complete questionnaires at baseline, 1 month, 3 months, and 6 months.

INTERVENTIONS:
Behavioral: Peer Network Counseling-txt — 4-week text counseling program
  Other Names: PNC-txt
  Arms: Intervention

SUMMARY:
The purpose of this study is to test a text-delivered counseling program to stop or reduce cannabis use among young adults (ages 18 to 25).

DETAILED DESCRIPTION:
After being informed about the study and potential risks, participants will complete online screening assessments. Those who are determined to be eligible via online screening will complete a urine drug screen to confirm eligibility. Once eligibility is confirmed, participants will be randomized either to the intervention group or to the wait-list control group. Those who are randomized to the intervention group will receive the 4-week text intervention via smartphone and complete assessments (including urine drug screens) at baseline, 1 month, 3 months, and 6 months. Those who are randomized to the wait-list control group will only complete the assessments (including urine drug screens) at baseline, 1 month, 3 months, and 6 months. Participants who are initially assigned to the wait-list control group can choose to receive the text intervention once their 6-month participation is complete.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 25 years old.
2. use of cannabis three or more days during a typical week.
3. a score of at least eight on the Cannabis Use Disorder Identification Test-Revised
4. a urine specimen positive for cannabis metabolites.
5. a score of at least two on the Mini International Neuropsychiatric Interview: Version 7.0.2 for DSM-V, Substance Use Disorder
6. must live in Tennessee or Colorado

Exclusion Criteria:

1. substance abuse treatment during the past three months.
2. lack of access to a text-capable phone.
3. unable or unwilling to commit to six months of follow-up.
4. not fluent in English.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1077 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2025-01-08 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Tetrahydrocannabinol (Delta-9-THC-COOH) levels | Baseline, 1 month, 3 months, 6 months
  Urine THC levels (50ng/mL, 100ng/mL, 200ng/mL, 300ng/mL) will provide a biological measure for current cannabis use.
Change in Past 30-Day Cannabis Use | Baseline, 1 month, 3 months, 6 months
  Past-30-day substance use (cannabis, alcohol, tobacco, other drugs) and consequences are measured using the Alcohol, Smoking and Substance Involvement Screening Test

SECONDARY OUTCOMES:
Change in Environmental Risk Assessment | Baseline, 1 month, 3 months, 6 months
  Participants will report using the Ecological Momentary Assessment reporting about Craving (0=none-10= intense), Cannabis Use (0=none-10= a lot), Mood (0=very good-10= very depressed), and Stress (0=no stress-10 = very stressed) on a 10 point scale for each item
Change in Young Adult Social Network Assessment | Baseline, 1 month, 3 months, 6 months
  Participants report information on each their 3 closest friends, representing their egocentric network. Individual friend scores are totaled based on all 8 risky and prosocial items (2-9). Thus, each peer's score has a potential range from -32 to 32, with greater scores indicating a healthier relationship. The total peer network health scores is based on the sum of all 24 risky and prosocial items across all three friends. Assuming three peers per participant, total network quality scores may range from -96 to 96, with lower scores indicating greater network risk and higher scores indicating greater network protection.
Cost Measures | 6 months
  Cost of intervention implementation will be compared to typical treatment cost for cannabis use disorder

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mason, Ph.D., Principal Investigator — University of Tennessee, Knoxville; J. Douglas Coatsworth, Ph.D., Principal Investigator — University of Tennessee, Knoxville
Locations (2):
- United States (2):
  - Colorado State University, Fort Collins, Colorado
  - University of Tennessee Knoxvile, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zaharakis N, Coatsworth JD, Riggs NR, Radford A, Rayburn S, Mennis J, Russell MA, Brown A, Mason MJ. Treating young adult cannabis use disorder with text message-delivered peer network counseling. Contemp Clin Trials. 2024 Sep;144:107635. doi: 10.1016/j.cct.2024.107635. Epub 2024 Jul 15. PMID 39019156